CLINICAL TRIAL: NCT00761384
Title: A Prospective Study With Individually Adjusted High Dose 90Y-Ibritumomab Tiuxetan Treatment With Peripheral Blood Stem Cells Support to Improve Outcome for Patients With Refractory/Recurrent B-cell Lymphoma, Stage II-IV
Brief Title: High Dose, Absorbed Dose Adjusted 90Y-ibritumomab With Peripheral Blood Stem Cells (PBSC) Support in B-cell Lymphoma
Acronym: HITT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6th radioimmunotherapy prot.; EudraCT number: 2007-002762-35
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2015-04

CONDITIONS: B-cell Lymphoma
Keywords: B-cell lymphoma; Refractory; Recurrent; 90Y-ibritumomab; Stem cells support; Dosimetry study
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 90Y-ibritumomab (Experimental): 90Y-ibritumomab given with stem cells support, based on absorbed dose escalation to the liver. Absorbed dose escalation starts at 12 Gy and is capped at 36 Gy to the liver.
  Interventions: Drug: 90Y-ibritumomab

INTERVENTIONS:
Drug: 90Y-ibritumomab — 90Y-ibritumomab given with stem cells support, based on absorbed dose escalation to the liver. Absorbed dose escalation starts at 12 Gy and is capped at 36 Gy to the liver.

SUMMARY:
90Y-ibritumomab given with stem cells support, based on absorbed dose escalation to the liver. Absorbed dose escalation starts at 12 Gy and is capped at 36 Gy to the liver.

ELIGIBILITY:
Inclusion Criteria:

* Written informed concent
* Age at least 18 years
* WHO Performance status 0-3
* Histologically verified B-cell lymphoma
* Diffuse large B-cell lymphoma and follicular grade III, failing an anthracycline containing regimen and patients not found suitable for a second line chemotherapy consolidated by high dose chemotherapy (HDCT) with stem cell support or radiotherapy
* Transformed B-cell lymphoma, failing first line therapy and not suitable for high dose chemotherapy (HDCT) or with a history of HDCT with stem cell support
* Follicular lymphoma grade II and I, and other indolent lymphomas must have failed second line treatment.
* One of these treatments must have contained chemotherapy and rituximab, the latter either together with chemotherapy or as maintenance.
* The lymphoma must require treatment, Mantle cell lymphoma, failing first line treatment,treatment required
* Measurable disease and the tumor burden must be acceptable according to the investigator
* Radiological studies must be performed and a unilateral bone marrow biopsy within 4 weeks before start of treatment
* Bone marrow reserve likely to give a harvest of at least 2x10 6 peripheral CD34+ stemcells or the existence of such a harvest or a corresponding central harvest
* Total bilirubin should not exceed 40 micromole/L
* A GFR as measured by Cystatin C of 50 ml/min
* HIV, Hepatitis B and C status known
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Known or clinical evidence of CNS involvement
* Bone marrow involvement at harvest as measured by biopsy and flow cytometry
* Subjects with prior radiation to a field that includes over or equal 25% of their red marrow, liver or lung or to both kidneys
* Prior chemotherapy or radiotherapy within 4 weeks
* Subjects who are pregnant or nursing
* Pulmonary involvement, that is not negligible at the discretion of the investigator
* Liver involvement of lymphoma
* History of hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Maximal tolerable dose (MTD) absorbed dose to the liver, safety and time to treatment failure (TTF) | 5 years

SECONDARY OUTCOMES:
Overall response (OR), complete response (CR), their duration, absorbed dose to normal organ and tumours, relapse pattern, the effect of radioimmunotherapy (RIT) in its own right as assessed by positron emission tomography (PET) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ola Lindén, MD, Principal Investigator — Lund University Hospital
Locations (1):
- Lund University Hospital, Lund, Sweden